CLINICAL TRIAL: NCT00497822
Title: To Study the Effect of Exercise Training in Term of Aerobic Exercise for 3 Months, on the Physical, Cognitive and Affective Function in Dementia Subjects
Brief Title: A Randomized Controlled Trial on the Effect of Exercise on Physical, Cognitive and Affective Function in Dementia Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KW/EX05-090; HARECCTR0500054
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Dementia
Keywords: Dementia
MeSH Terms: conditions — Dementia

INTERVENTIONS:
Procedure: Aerobic exercise training

SUMMARY:
Studies have shown conflicting results of the effect of exercise on dementia patients.

The aim of this study is to examine the role of physical activity on the risk of cognitive impairment and dementia in older persons.

To promote the benefits of aerobic exercise on dementia patients and encourage exercise prescription in the management of dementia subjects.

ELIGIBILITY:
Inclusion Criteria:

* MMSE<26
* Age >60
* Community dwelling and ambulatory
* Have a caregiver that is willing to participate and escort patient to hospital for training and assessment

Exclusion Criteria:

* MMSE<10
* live in old age home
* poor mobility, unable to attend exercise training
* no carer to bring patient to attend hospital training

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-01; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Physical function measurement using SF-12 | every 3 months for 1 year
Affective function measurement by Cornell depression score | every 3 months for 1 year
Cognitive function by MMSE and ADAS-cog | every 3 months for 1 year

SECONDARY OUTCOMES:
6 minutes walk, functional reach, Berg balance scale | every 3 months for 1 year
Carer stress scale | every 3 months for 1 year
No. of fall/restricted activity days/time spend in exercise or walking | every 3 months for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Doris KY Miu, Dr, Principal Investigator — Department of Medicine and Geriatrics, Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, China